CLINICAL TRIAL: NCT00594607
Title: A Comparing Study of Nephral 400 ST and Fx8 Dialysis Membranes on Coagulation During Hemodialysis
Brief Title: Effect of Nephral 400 ST Dialysis Membrane on Coagulation in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Rikshospitalet University Hospital (Other)
Responsible Party: Solbjørg Sagedal, MD, PhD, Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: S-04147; NSD-data services 11056
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2008-05

CONDITIONS: Extracorporeal Clotting During Hemodialysis
Keywords: clotting; hemodialysis; anticoagulation; bleeding risk
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: AN69ST (Active Comparator): Hemodialysis sessions with use of the dialysis filter AN69ST.
  Interventions: Device: AN69ST dialysis membrane
- 2:Fx8 (Active Comparator): Hemodialysis sessions with use of the dialysis filter Fx8
  Interventions: Device: Fx8 (Fresenius)

INTERVENTIONS:
Device: AN69ST dialysis membrane — AN69ST is the filter that the blood goes through during hemodialysis
  Arms: 1: AN69ST
Device: Fx8 (Fresenius) — Polysulphone dialysis membrane
  Arms: 2:Fx8

SUMMARY:
The purpose of this study is to investigate whether the dialysis filter AN69ST (Nephral 400 ST Dialysis Membrane) induces less clotting during hemodialysis than a conventional polysulphone filter. Our hypothesis is that the two filters induce the same degree of clotting.

DETAILED DESCRIPTION:
Six consecutive hemodialysis (HD) sessions are evaluated per patient, altogether 10 - 12 stable HD patients (or at least 48 HD sessions altogether). During these six sessions, AN69ST and Fx8 are used on alternate days. Dalteparin is given intravenously as a single bolus dose at start of HD (50% of the conventional dose). Clinical clotting is evaluated visually each hour of HD after blood draining of the venous air trap: 1=no clot, 2=a fibrinous ring, 3=a clot <1 cm, 4=a clot >1 cm and 5=coagulated system (stop in HD).

Blood specimens are taken at start and after each hour of HD. Markers of coagulation (prothrombin 1+2) and of platelets (beta-thromboglobulin) are evaluated as well as anti FXa-activity.

The two filters are going to be compared statistically with respect to the degree of clinical clotting and of intravascular coagulation and platelets activation.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 18 years or more having been in chronic HD for at least 1 month
* dialysis time at least 4 hours 3 times per week
* blood flow at least 200 ml/min
* Fragmin dose unchanged the last week before study start
* Fragmin given intravenously as one single dose at HD start
* Haemoglobin >= 11.0 g/dL and stable +/- 20% the last week before study start
* erythropoietin and iron dose unchanged the last week before study start
* written and orally informed consent given by the patient

Exclusion Criteria:

* treatment with acetylsalicylic acid (ASA)
* use of Warfarin or another oral anticoagulant
* clinical signs of infection
* disseminated malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Clinical clotting in the air trap | 14 days (6 consecutive HD sessions)

SECONDARY OUTCOMES:
Intravascular coagulation and platelet activation | 14 days (6 HD sessions)

CONTACTS AND LOCATIONS:
Overall Officials: Solbjørg Sagedal, PhD, MD, Principal Investigator — Department of Nephrology, Ullevål University hospital, 0407 Oslo; Anders Hartmann, PhD, MD, Study Director — Department of Internal medicine, Rikshospitalet University Hospital, 0027 Oslo; Solbjørg Sagedal, PhD, MD, Study Chair — department of Nephrology, Ullevål University Hospital, Oslo
Locations (1):
- Department of Nephrology, Ullevål University Hospital, Oslo, Norway